CLINICAL TRIAL: NCT02159183
Title: A Controlled Clinical Pilot Study to Assess Soft Tissue Reaction at the Crestal Part of a Dental Implant With ESTA Surface
Brief Title: Controlled Pilot Study to Assess Soft Tissue Reaction at the Crestal Part of a Dental Implant With ESTA Surface
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 5-Y FUP will not result in new perception, no diff. between groups at 1+3y FUP
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR 01/11
Record Dates: First submitted 2014-06-03; First posted 2014-06-09 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Teeth Loss
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Plus ESTA STL Roxolid implant (Experimental): This arm will receive the Straumann Soft Tissue Level Standard Plus Implant Ø 4.1 mm Regular Neck, SLActive® Roxolid, with a modified surface of the neck (ESTA).
  Interventions: Device: Standard Plus ESTA STL Roxolid implant
- Standard Plus STL implant (Active Comparator): This arm will receive the Straumann Soft Tissue Level Standard Plus Implant Ø4.1mm Regular Neck,SLActive® Titanium grade IV, with a machined surface of the neck.
  Interventions: Device: Standard Plus STL implant

INTERVENTIONS:
Device: Standard Plus ESTA STL Roxolid implant — The patient will receive a Straumann Soft Tissue Level Standard Plus Implant Ø 4.1 mm Regular Neck, SLActive® Roxolid, with a modified surface of the neck (ESTA). At 8-12 weeks after insertion, the implant will be loaded.
  Arms: Standard Plus ESTA STL Roxolid implant
Device: Standard Plus STL implant — The patient will receive a Straumann Soft Tissue Level Standard Plus Implant Ø4.1mm Regular Neck,SLActive® Titanium grade IV, with a machined surface of the neck. At 8-12 weeks after insertion, the implant will be loaded.
  Arms: Standard Plus STL implant

SUMMARY:
This study will investigate the effect on the soft tissue that is in contact with a dental implant with a modified surface of the neck (the part of the implant that is above the bone and in contact with the soft gum tissue).

DETAILED DESCRIPTION:
This is a prospective, controlled, randomised clinical pilot study with parallel groups and blinded subject.

The design has been chosen to obtain data to base a sample size calculation for future studies on by comparing the degree of mucosal inflammation of the mucosa in conjunction with the modified surface of the top of the test implant and the machined surface on the top of the control implant.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have voluntarily signed the informed consent form before any study related action
* Males and females must be at least 18 years of age and not more than 80 years old.
* Partially edentulous in posterior (position 3-7) maxilla or mandible with implants planned for single crowns in an area with a healed extraction socket.
* Adequate bone quality and quantity at the implant site to permit the insertion of a Straumann Soft Tissue Level implant of 4.1mm diameter without augmentation (at least 1mm bone buccally and lingually/palatal)

Exclusion Criteria:

* Oral surgery contraindicated according to the judgement of the investigator (should be explained in the CRF)
* Local inflammation, including untreated periodontitis
* Patients with inadequate oral hygiene or unmotivated for adequate home care. Full mouth plaque index > 25% at time of surgery
* Presence of conditions requiring chronic routine prophylactic use of antibiotics (e.g., history of rheumatic heart disease, bacterial endocarditis, cardiac valvular anomalies, prosthetic joint replacements)
* Major systemic diseases
* Medical conditions requiring prolonged use of steroids
* Current pregnancy or breastfeeding women
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene
* Use of any investigational drug or device within the 90 day period immediately prior to implant surgery on study day 0
* Alcoholism or chronically drug abuse
* Smokers; more than 10 cigarettes per day
* Immuno-compromised patients
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, or unreliability.

Secondary Exclusion Criteria:

* GBR procedures at or adjacent to the planned study site
* Lack of primary stability of the dental implant at site of interest (e.g., rotational movement of the implant at a minimum of 15 Ncm torque at connection of the healing abutment, or tactile mobility)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2016-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anton Sculean, Prof. Dr., Principal Investigator — Universität Bern, Klinik für Parodontologie
Locations (4):
- Switzerland (4):
  - University of Bern, Bern
  - University of Geneva, Geneva
  - Private Practice, Langenthal
  - Ardentis Clinique Dentaire, Lausanne

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Analysis After the 36 Months Follow-up
Arm/Group | Standard Plus ESTA STL Roxolid Implant | Standard Plus STL Implant
Started | 22 | 21
Completed | 19 | 19
Not Completed | 3 | 2
Not completed — Protocol Violation | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Death | 0 | 1
Period: Analysis of Primary Endpoint (12 Mts)
Arm/Group | Standard Plus ESTA STL Roxolid Implant | Standard Plus STL Implant
Started | 22 | 21
Completed | 19 | 20
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Population: Number of participants randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Plus ESTA STL Roxolid Implant | Standard Plus STL Implant | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (13) | 56 (13) | 57 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 11 | 8 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  Switzerland: center "Bern/Switzerland" | 7 | 7 | 14
  Switzerland: center "Langenthal/Switzerland" | 7 | 6 | 13
  Switzerland: center "Geneva/Switzerland" | 5 | 5 | 10
  Switzerland: center "Lausanne/Switzerland" | 3 | 3 | 6
Full Mouth Bleeding on Probing (FMBoP) [Mean (Standard Deviation); unit: %] — Full mouth bleeding index on probing is an indicator for Oral Hygiene and is measured in percent [%].
  Percentage of total surfaces with bleeding = Number of surfaces with bleeding divided by the total number of tooth surfaces x 100
  % | 14.2 (6.0) | 13.3 (6.2) | 13.7 (6.0)
Full Mouth Plaque Index (FMPI) [Mean (Standard Deviation); unit: %] — Full mouth plaque index (FMPI) is an indicator for Oral Hygiene and is measured in percent [%].
  Percentage of total surfaces with plaque = number of surfaces with plaque divided by the total number of tooth surfaces x 100.
  % | 18.7 (3.8) | 15.9 (5.5) | 17.3 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Sulcus Bleeding Index (According to Mombelli et al 1987)
Description: The primary endpoint is the difference of Sulcus Bleeding Index (according to Mombelli et al 1987) between baseline (final loading) and 12 months.
  The inflammatory status of the mucosa will be evaluated by means of a UNC 15 periodontal probe.
  0: No bleeding when a periodontal probe is passed along the peri-implant sulcus
  1. Isolated bleeding spots are recognizable
  2. Confluent bleeding line along the marginal mucosa
  3. Profound bleeding.
Time Frame: 12 months
Population: per protocol analysis
Measure: Count of Units; unit: sites on teeth
Units Other Than Participants: sites on teeth
Arm/Group | Standard Plus ESTA STL Roxolid Implant | Standard Plus STL Implant
Number analyzed (Participants) | 19 | 20
Number analyzed (sites on teeth) | 76 | 80
sites on teeth
  confluent bleeding -> isolated bleeding | 1 | 0
  isolated bleeding --> no bleeding | 5 | 9
  isolated bleeding --> isolated bleeding | 2 | 3
  no bleeding -> no bleeding | 51 | 53
  no bleeding -> isolated bleeding | 16 | 14
  no bleeding -> confluent bleeding | 1 | 1

2. Secondary Outcome: Sulcus Bleeding Index (According to Mombelli et al 1987)
Description: The inflammatory status of the mucosa will be evaluated by means of a UNC 15 periodontal probe.
  0: No bleeding when a periodontal probe is passed along the peri-implant sulcus
  1. Isolated bleeding spots are recognizable
  2. Confluent bleeding line along the marginal mucosa
  3. Profound bleeding.
Time Frame: 3 years
Population: Per-Protocol Analysis
Measure: Number; unit: Sites on teeth
Units Other Than Participants: Sites on teeth
Arm/Group | Standard Plus ESTA STL Roxolid Implant | Standard Plus STL Implant
Number analyzed (Participants) | 19 | 19
Number analyzed (Sites on teeth) | 76 | 76
Sites on teeth
  No Bleeding | 59 | 60
  Bleeding | 17 | 16

3. Secondary Outcome: Soft Tissue Healing Evaluation
Description: Assessment of the wound healing by classifying the implantation site (normal or compromised healing).
Time Frame: 10 days and 12 weeks
Measure: Number; unit: participants
Arm/Group | Standard Plus ESTA STL Roxolid Implant | Standard Plus STL Implant
Number analyzed (Participants) | 22 | 21
participants
  normal healing, 10 days | 22 | 21
  normal healing, 12 weeks | 22 | 21

4. Secondary Outcome: Oral Hygiene
Description: Full mouth plaque index (FMPI) and full mouth bleeding on probing index (FMBoP) will be recorded as an indicator for the Oral Hygiene. The indexes are given in percent [%] calculated as the total numbers of surfaces with plaque or bleeding divided by the total number of teeth surfaces x100.
Time Frame: Screening, 6, 12, 36 months
Population: Per-protocol analysis. Missing data on some patients
Measure: Mean (Standard Deviation); unit: percentage of surfaces
Arm/Group | Standard Plus ESTA STL Roxolid Implant | Standard Plus STL Implant
Number analyzed (Participants) | 22 | 21
percentage of surfaces
  FMBoP, screening: number analyzed (Participants) | 19 | 19
  FMBoP, screening | 14 (6) | 15 (6)
  FMBoP, 6 Months: number analyzed (Participants) | 19 | 18
  FMBoP, 6 Months | 13 (6) | 11 (6)
  FMBoP, 1 year: number analyzed (Participants) | 19 | 19
  FMBoP, 1 year | 14 (5) | 11 (5)
  FMBoP, 3 years: number analyzed (Participants) | 19 | 19
  FMBoP, 3 years | 16 (8) | 15 (7)
  FMPI, screening: number analyzed (Participants) | 19 | 19
  FMPI, screening | 19 (4) | 16 (6)
  FMPI, 6 Months: number analyzed (Participants) | 19 | 17
  FMPI, 6 Months | 14 (6) | 14 (6)
  FMPI, 1 year: number analyzed (Participants) | 19 | 19
  FMPI, 1 year | 16 (5) | 14 (4)
  FMPI, 3 years: number analyzed (Participants) | 19 | 19
  FMPI, 3 years | 17 (8) | 18 (8)

5. Secondary Outcome: Recession of Gingival Margin Buccally and Lingually/Palatal
Description: The recession of the gingival margin will be measured (distance from the gingival margin to the crown/implant margin) by using an UNC 15 periodontal probe. Changes in (averaged) recession at the follow-up visits 12+36 months compared to baseline visit ( final loading ) are displayed
Time Frame: 1 and 3 years
Population: Per protocol Analysis. Missing data of some patients.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Standard Plus ESTA STL Roxolid Implant | Standard Plus STL Implant
Number analyzed (Participants) | 22 | 21
mm
  Difference in recession 1 yr to final loading: number analyzed (Participants) | 19 | 19
  Difference in recession 1 yr to final loading | -0.5 (0.9) | -0.6 (1.1)
  Difference in recession 3 yr to final loading: number analyzed (Participants) | 19 | 19
  Difference in recession 3 yr to final loading | -0.5 (1.1) | -0.7 (1.1)

6. Secondary Outcome: Probing Pocket Depth (PPD)
Description: The PPD will be measured from the mucosal margin to the bottom of the periimplant pocket by means of an UNC 15 probe.
  Probing pocket depth (mm) - average over buccal, palatal, distal and mesial measurements.
Time Frame: 6 months, 1 and 3 years
Population: Per-Protocol Analysis. Missing data of some of the patients
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Standard Plus ESTA STL Roxolid Implant | Standard Plus STL Implant
Number analyzed (Participants) | 22 | 21
mm
  PPD average, 6 Months: number analyzed (Participants) | 19 | 18
  PPD average, 6 Months | 3.0 (0.5) | 2.8 (0.4)
  PPD average, 1 year: number analyzed (Participants) | 19 | 19
  PPD average, 1 year | 3.1 (0.6) | 2.9 (0.6)
  PPD average, 3 years: number analyzed (Participants) | 19 | 19
  PPD average, 3 years | 3.2 (0.8) | 3.0 (0.6)

7. Secondary Outcome: Clinical Attachment Level (CAL)
Description: The CAL will be measured from the crown margin to the bottom of the periimplant pocket by means of an UNC 15 probe.
  Clinical attachment level (mm) - average over buccal, palatal, distal and mesial measurements
Time Frame: 6 months, 1 and 3 years
Population: Per-Protocol Analysis. Missing data of some of the patients
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Standard Plus ESTA STL Roxolid Implant | Standard Plus STL Implant
Number analyzed (Participants) | 22 | 21
mm
  CAL average, 6 months: number analyzed (Participants) | 19 | 18
  CAL average, 6 months | 1.9 (0.5) | 1.8 (0.7)
  CAL average, 1 year: number analyzed (Participants) | 19 | 19
  CAL average, 1 year | 2.0 (0.7) | 2.1 (0.7)
  CAL average, 3 years: number analyzed (Participants) | 19 | 19
  CAL average, 3 years | 1.9 (0.7) | 2.1 (0.7)

8. Secondary Outcome: Bone Crest Levels. Bone Levels (mm) - Average Over Mesial+Distal Measurements
Description: Periapical radiographs are used to measure changes in mesial and distal bone crest levels (of the implant) from baseline (final loading) to one (1) year and three (3) years, respectively.
  The parameter derives from the subtraction of mesial and distal bone level linear x-ray measurements. The distance between the alveolar bone at the level of the first radiographic bone contact with the implant surface, and the shoulder of the implant will be measured to the closest 0.1mm at the mesial and distal surfaces of all implants on digitized standardized periapical x-rays using an image analysis computer programme. Bone levels are averaged over mesial+distal measurements. Since bone levels were measured from the implant shoulder, an increase in bone level over time corresponds to bone loss.
Time Frame: 1 and 3 years
Population: Per-Protocol Analysis. Missing data of some of the patients
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Standard Plus ESTA STL Roxolid Implant | Standard Plus STL Implant
Number analyzed (Participants) | 22 | 21
mm
  Bone level change from 1 year to baseline: number analyzed (Participants) | 18 | 19
  Bone level change from 1 year to baseline | 0.24 (0.59) | 0.14 (0.3)
  Bone level change from 3 years to baseline: number analyzed (Participants) | 18 | 19
  Bone level change from 3 years to baseline | 0.33 (0.69) | 0.12 (0.3)

9. Secondary Outcome: Dental Implant Success and Implant Loss
Description: The implant success will be defined according to Buser et al 1990. Overall evaluation of implant success.
Time Frame: 3 years
Population: Intention to Treat (ITT) Analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Plus ESTA STL Roxolid Implant | Standard Plus STL Implant
Number analyzed (Participants) | 22 | 21
Participants
  Patient with implant loss, 3 years | 1 | 0
  Successful after 3 years | 19 | 18

10. Secondary Outcome: Adverse Events
Description: All subjects are monitored continuously for adverse event.
Time Frame: up to 3 years
Population: ITT Analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Plus ESTA STL Roxolid Implant | Standard Plus STL Implant
Number analyzed (Participants) | 22 | 21
Participants | 11 | 11

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Standard Plus ESTA STL Roxolid Implant | Standard Plus STL Implant
All-Cause Mortality (participants affected / at risk) | 0/22 | 1/21
Serious Adverse Events (participants affected / at risk) | 1/22 | 2/21
Other Adverse Events (participants affected / at risk) | 10/22 | 9/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Plus ESTA STL Roxolid Implant (N=22) | Standard Plus STL Implant (N=21)
Kneeoperation (Musculoskeletal and connective tissue disorders) | 1 | 0
Ablation of a cyste in the femur (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Death (Cardiac disorders) | 0 | 1 — Patient died of heart attack
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Plus ESTA STL Roxolid Implant (N=22) | Standard Plus STL Implant (N=21)
Tooth related events (General disorders) | 2 (4) | 4 (5)
Implant related events (Surgical and medical procedures) | 4 (4) | 1 (1)
Prosthetic related events (Surgical and medical procedures) | 3 (3) | 3 (4)
Non-related clinical conditions (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days